CLINICAL TRIAL: NCT00338156
Title: Assessment of the Relationship Between Collagen Turnover, Left Ventricular Remodelling and Myocardial Scarring Assessed by Cardiac Magnetic Resonance and Neurohumoral Activation in Patients With Previous Myocardial Infarction
Brief Title: Observational Study of the Remodelling Process Following Myocardial Infarct
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); Amersham Buchler, GmbH & Co KG (Industry)
Responsible Party: Sponsor
Other Study IDs: StaHF461302; Helse Vest 911017 (Other Grant/Funding Number: Helse Vest RHF)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Heart Failure; Myocardial Infarct
Keywords: Left Ventricle Remodelling; Collagen markers; Neurohormones; Cardiac MRI
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess the relationship between collagen turnover, neurohormonal activation, scarring and left ventricle remodelling in patients 3 years following a myocardial infarction.

DETAILED DESCRIPTION:
A multinational trial compared losartan vs. captopril in 5477 postinfarction patients with symptoms of heart failure and/or evidence of left ventricular dysfunction. The trial was terminated in 2002 and the results of the main trial have been published. In this trial, a collagen and neurohumoral substudy was performed to assess the importance of collagen turnover in this population. A total of 235 patients were included from 18 centres. Blood was taken at randomisation, 1 month, 1 year and 2 years.

The present study will recruit surviving patients among the 119 individuals that were randomised to the neurohumoral substudy at the Stavanger University Hospital. The study will assess the relationship between collagen turnover, neurohormonal activation, scarring and left ventricle remodelling in these patients about 3 years following the index myocardial infarction.

The data collected at the 3-year follow-up visit will be compared to data from the initial study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the previous neurohormonal substudy of the OPTIMAAL trial
* Willingness to participate in the present study and ability to understand and sign the written informed consent

Exclusion Criteria:

* Myocardial infarction within 3 months of visit 1.
* Significant primary valve disease, confirmed by ECHO cardiography,
* Autoimmune disease likely to cause an increase in collagen turnover
* Active cancer disease
* Immunosuppressive treatment,
* Significantly reduced liver function
* Contraindications for performing a cardiac MRI scan (including claustrophobia, implanted ferromagnetic devices or known allergic reactions to Omniscan™).
* Inability to cooperate during the 1 month follow up period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with risk of heart failure secondary to myocardial infarct.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dickstein, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway